CLINICAL TRIAL: NCT00988156
Title: Efficacy and Safety Study of Eslicarbazepine Acetate (BIA 2 093) as Adjunctive Therapy for Refractory Partial Seizures in Children
Brief Title: Eslicarbazepine Acetate (BIA 2 093) as Therapy for Refractory Partial Seizures in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-2093-305; 2007-001887-55 (EudraCT Number)
Record Dates: First submitted 2009-10-01; First posted 2009-10-02 (Estimated); Results first posted 2014-07-17 (Estimated); Last update posted 2018-11-13 (Actual); Status verified 2018-10

CONDITIONS: Partial Epilepsy in Children and Adolescents
Keywords: Epilepsy; Partial; Refractory; Children; Adolescents; Adjunctive; Randomised; Double-blind; Placebo-controlled; Parallel-group
MeSH Terms: conditions — Epilepsy | interventions — eslicarbazepine acetate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eslicarbazepine acetate (Active Comparator): To receive Eslicarbazepine acetate in addition to concomitant therapy
  Interventions: Drug: Eslicarbazepine acetate (BIA 2-093)
- Placebo (Placebo Comparator): To receive placebo in addition to concomitant therapy
  Interventions: Drug: Eslicarbazepine acetate

INTERVENTIONS:
Drug: Eslicarbazepine acetate (BIA 2-093) — Part I - 8-week observational baseline period followed by a 6-week double-blind titration period, a 12-week double-blind maintenance period, a double-blind tapering-off period, and a 4-week observational period.
  The recommended target dose of double-blind study treatment will be 20mg/kg/day.
  Part II: At the end of part I, there is an option to enter a long-term open-label extension period to receive Eslicarbazepine acetate for 1 year.
  Other Names: BIA 2093
  Arms: Eslicarbazepine acetate
Drug: Eslicarbazepine acetate — Part I: 8-week observational baseline period followed by a 6-week double-blind titration period, a 12-week double-blind maintenance period, a double-blind tapering-off period, and a 4-week observational period.
  Part II: At the end of part I, there is an option to enter a long-term open-label extension period to receive Eslicarbazepine acetate for 1 year.
  Other Names: BIA 2093
  Arms: Placebo

SUMMARY:
The purpose of this study is to examine the efficacy and safety of Eslicarbazepine acetate (BIA 2-093) when given with other anti-epileptic drugs to treat children with partial seizures whose condition has not been controlled by other drug treatments.

DETAILED DESCRIPTION:
Partial epilepsy, the commonest form of epilepsy, is a difficult condition to treat with many patients continuing to have symptoms despite trying several medications. Lack of efficacy and adverse effects are commonly associated with current anti-epileptic drugs.

This study will examine the efficacy in addition to safety and tolerability of a new anti-epileptic drug, Eslicarbazepine acetate (BIA 2-093), as an adjunctive therapy for refractory partial seizures in children.

The primary analysis variables are:

* The responder rate (the proportion of patients with at least a 50% reduction in standardised seizure frequency)
* The relative reduction in standardised seizure frequency

ELIGIBILITY:
Inclusion Criteria:

* girls of child-bearing potential have to follow reliable and medically acceptable contraceptive method throughout the study
* diagnosis of epilepsy for at least 6 months prior to enrolment
* at least 4 partial-onset seizures in the last month prior to enrolment despite stable therapy with adequate dosage of 1 or 2 AEDs
* at least 4 partial-onset seizures during each 4-week interval of the 8-week baseline period
* previous treatment with three or more AEDs, in their maximum tolerated doses, for at least one month, without seizure control
* current treatment with 1 or 2 AEDs (any except oxcarbazepine); if present, vagus nerve stimulation is considered an AED
* stable dose regimen of AEDs during the 8-week baseline period
* cooperation and willingness to complete all aspects of the study, including hospitalisation if required
* written informed consent to participate in the study in accordance with local legislation

Exclusion Criteria:

* primarily generalised seizures
* baseline seizure frequency substantially different from usual seizure frequency
* known progressive neurological disorders
* history of status epilepticus within the 3 months prior to enrolment
* seizures of non-epileptic origin
* Lennon-Gastaut
* West syndrome
* Major psychiatric disorders
* Previous treatment any study with Eslicarbazepine acetate

Ages: 2 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 304 (Actual)
Dates: Start 2007-12-07 (Actual); Primary Completion 2012-08-20 (Actual); Study Completion 2017-08-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (91):
- Austria (2):
  - Ambulanz für Neuropädiatrie und Entwicklungsdiagnostik, Med. Univ. Graz, Graz
  - Universitätsklinik für Kinder- und Jugendheilkunde, Klinische Abteilung für allg. Pädiatrie, AKH Wien, Vienna
- Bosnia and Herzegovina (2):
  - Clinical Centre Banja Luka Pediatric Clinic Department of Neurology, Banja Luka
  - Clinical Center University of Sarajevo Pediatric Clinic Neuropediatrics Department, Sarajevo
- Croatia (3):
  - Clinical hospital Osjek Pediatric clinic, neuropediatric department, Osijek
  - Clinic for Children Diseases Zagreb, Zagreb
  - Clinic for Sick Children "Dr. Sabol", Zagreb
- Czechia (5):
  - Clinic of the Child Neurology, FN Brno, Brno
  - Neurology Policlinic, Hradec Králové
  - Child Neurology Clinic of the DNsP Ostrava, Ostrava
  - Department of the Child Neurology FTN, Prague
  - Children Neurology Clinic, University Hospital Motol, Prague
- France (5):
  - CHU Hopital Nord, Amiens
  - Hopital Pédiatrique Enfants, Bordeaux
  - Hopital Enfants de la Timone, Marseille
  - Université Paris Descartes, Hopital Necker-Enfants Malades, Département de Neuropédiatrie, Paris
  - Hopital des Enfants, Toulouse
- Germany (2):
  - Epilepsiezentrum Kehl-Kork Kinderklinik Anfallsambulanz für Kinder und jugendliche, Kehl-Kork
  - Familienpraxis Oggersheim, Ludwigshafen
- Hungary (3):
  - Budai Gyermekkórház, Buda Children's Hospital and Outpatient Clinic, Budapest
  - Children Neurology Dept., Borsod-Abaúj-Zemplén Megyei Kórház és Egyetemi Oktató Kórház, Miskolc
  - Pécsi Tudományegyetem AOK Gyermekklinika, Pécs
- Italy (7):
  - A.O.U. di Cagliari Clinica di neurologia infantile, Cagliari
  - Ospedale Petiatrico IRCCS, Genova
  - A. O. C. "Poma", Mantova
  - Fondazione Istituto Neurologico Casimiro Mondino, Pavia
  - Dipartimento di Neuroscienze, Unità Operativa di Neurologia Ospedale Bambin Gesù, Rome
  - Azienda Ospedaliera Universitaria Senese Ospedale Santa Maria alle Scotte Dipartimento materno infantile Struttura Complessa di Pediatria, Siena
  - Servizio di Neuropsichiatria Infantile Policlinico "G.B. Rossi" Borgo Roma, Verona
- Malaysia (2):
  - Hospital Raja Perempuan Zainab II - Jabatan Paediatrik, Kelantan, Kelantan
  - University Putra Malaysia/Hospital Serdang - Department of Paediatrics, Faculty of Medicine and Health Sciences, Kuala Selangor, Selangor
- IMSP Centrul National Stiintifico-Practic Medicina de Urgenta, Chishinau, Moldova
- Philippines (5):
  - Cebu Davao Doctors Hospital, Cebu City, Cebu
  - Perpetual Succour Hospital - Neuroscience Center, 7/F SPC Medical Specialty Center, Cebu City, Cebu
  - Davao Doctor's Hospital, Davao City, Davao Del Sur
  - Manila Doctors Hospital - Child Nueroscience Center, Ermita, Manila
  - Jose R. Reyes Memorial Medical Center - 5th Floor, Training and Research Office, Jose Reyes Memorial Hospital, Santa Cruz, Manila
- Poland (7):
  - SAMODZIELNY PUBLICZNY SZPITAL KLINICZNY NR 6 ŚLĄSKIEJ AKADEMII MEDYCZNEJ W KATOWICACH GÓRNOŚLĄSKIE CENTRUM ZDROWIA DZIECKA I MATKI IM. JANA PAWŁA II Klinika Pediatrii i Neurologii Wieku Rozwojowego, Katowice
  - Instytut Neuromedica, Krakow
  - Krakowski Szpital, Specjalistyczny Im. Jana Pawła Ii W Krakowie, Krakow
  - WOJEWÓDZKI SPECJALISTYCZNY SZPITAL DZIECIĘCY im. ŚW. LUDWIKA W KRAKOWIE, Krakow
  - Instytut "Centrum Zdrowia Matki Polki" Klinika Neurologii, Lodz
  - AKADEMIA MEDYCZNA im. Karola Marcinkowskiego w Poznaniu Katedra I Klinika Neurologii Wieku Rozwojowego, Poznan
  - Przychodnia NEUROSPHERA, Warsaw
- Portugal (7):
  - Hospital Pediátrico de Coimbra, Coimbra
  - Hospital Dona Estefânia, Lisbon
  - Hospital Francisco Xavier, Lisbon
  - Hospital Santa Maria, Lisbon
  - Hospital Pedro Hispano, Matosinhos Municipality
  - Hospital Geral de Santo António, Porto
  - Hospital Maria Pia, Porto
- Romania (3):
  - Clinica de Neurologie Peciatrica, Spitalul "Alexandru Obregia", Bucharest
  - Clinical Hospital for children, Paediatric Neurology clinic, Cluj-Napoca
  - Spitalul Clinic de Urgenta pentru copii Luis Turcanu, Clinica de Psihiatrie si Neurologie pentru copii si adolescenti, Timișoara
- Russia (6):
  - Pediatric Scientific-practical Center of cranio-facial surgery and neurology, Moscow
  - Research Center of Children Health of RAMS, Moscow
  - Moscow Research Institute of Pediatrics and Pediatric Surgery of Rosmedtechnology, Moscow
  - Nizhny Novgorod State Medical Academy Pediatric City Clinical Hospital No. 1, Nizhny Novgorod
  - Neurological Department, Voronezh Regional Pediatric Clinical Hospital No. 1, Voronezh
  - Department of Neurolog, Regional Pediatric Clinical Hospital No. 1 Ekaterinburg, Yekaterinburg
- Serbia (4):
  - Child Neurology Service, Institute of Mother and Child Healthcare of Serbia "Dr. Vukan Cupic", Belgrade
  - Clinic of Neurology and Psychiatry for Children and Youth, Belgrade
  - Clinical Centre Nis, Clinic of Children Internal Diseases, Child Neurology Department, Niš
  - Children Neurology Dept., Institute of Child- and Adolescent Health Care of Vojvodina, Novi Sad
- Slovakia (4):
  - Child Epileptology Out-patient, Dolný Kubín
  - Neurologická ambulancia, Dubnica nad Váhom
  - Neurologická ambulancia, Hlohovec
  - Tempus, s.r.o.Child Epileptology Ambulance, Liptovský Mikuláš
- Spain (8):
  - IMAS Hospital del Mar - Servicio de Pediatria, Barcelona
  - Hospital Vall Hebron, Barcelona
  - Hospital Sant Joan de Déu, Dep. Neuropediatría, Esplugues de Llobregat
  - Hospital Materno Infantil Virgen de las Nieves, Granada
  - Hospital Clínico San Carlos, Servicio de Neurología Pediátrica, Madrid
  - Hospital Son Dureta Dep. Neuropediatría, Palma de Mallorca
  - Hospital Son Dureta, Dep. Neuropediatría, Palma de Mallorca
  - Hospital Universitario Miguel Servet, Zaragoza
- Taiwan (2):
  - National Taiwan University Hospital - Department of Paediatrics, Taipei
  - Taipei Veterans General Hospital - Department of Paediatrics, Taipei
- Ukraine (4):
  - Pediatric Clinical Hospital No. 5, Department of Pediatric Neurology, Dnipro
  - Institute of Neurology, Psychiatry and Narcology, AMS of Ukraine Acad., Kharkiv
  - Ukrainian Medical Rehabilitation Centre for Children with Organic Disorders of Nervous System, Kiev
  - Hospital pediatrics of Odessa State Medical University Odessa, Odesa
- United Kingdom (9):
  - Birmingham Children's Hospital, Birmingham
  - Crawley Hospital, Crawley
  - Department of Paediatric, Clarendon Wing, Leeds General Infirmary, Leeds
  - The Royal London Hospital, London
  - St Georges Hospital, Child Development, London
  - Great Ormond Street Hospital, London
  - Royal Victoria Infirmary Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne
  - Queen's Hospital, Romford
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Mintz M, Pina-Garza JE, Wolf SM, McGoldrick PE, Jozwiak S, Grinnell T, Cantu D, Costa R, Moreira J, Li Y, Blum D. Safety and Tolerability of Adjunctive Eslicarbazepine Acetate in Pediatric Patients (Aged 4-17 Years) With Focal Seizures. J Child Neurol. 2020 Mar;35(4):265-273. doi: 10.1177/0883073819890997. Epub 2019 Dec 26. PMID 31878820
- See also: Sponsor Web page for Clinical Trials Transparency — https://www.bial.com/en/r_d.2/transparency.208/clinical_trials.209/eslicarbazepine_acetate.210.html
- See also: EU Clinical Trials Register: Clinical Trial Results — https://www.clinicaltrialsregister.eu/ctr-search/trial/2007-001887-55/results

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 73 clinical centres in 20 countries Date first patient enrolled: 07 Dec 2007. Date last patient completed the double-blind treatment period (Part I): 20 Aug 2012.
Groups:
- Placebo: Placebo matching placebo
- Esl (BIA 2-093): Eslicarbazepine acetate (Esl) (BIA 2-093) The study treatment was ESL. These treatments were provided as an oral suspension (50 mg/mL) and as white oblong tablets (200 mg).
Period: Overall Study
Arm/Group | Placebo | Esl (BIA 2-093)
Started | 149 | 155
Intention-to-Treat Set (ITT) | 129 | 134
Per Protocol Set (PP) | 101 | 97
Safety Set | 129 | 134
Completed | 132 | 135
Not Completed | 17 | 20

BASELINE CHARACTERISTICS:
Groups:
- Esl (BIA 2-093): Eslicarbazepine acetate (Esl) (BIA 2-093) The study treatment was ESL or matching placebo. These treatments were provided as an oral suspension (50 mg/mL) and as white oblong tablets (200 mg).
- Total: Total of all reporting groups
Arm/Group | Placebo | Esl (BIA 2-093) | Total
Number analyzed (Participants) | 129 | 134 | 263
Age, Customized [Number; unit: participants]
  2-6 years | 31 | 31 | 62
  7-11 years | 53 | 51 | 104
  12-18 years | 45 | 52 | 97
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 70 | 137
  Male | 62 | 64 | 126

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Seizure Frequency
Description: Relative reduction in the standardised 4-week seizure frequency from the baseline period to the 12-week maintenance period.
Time Frame: Baseline up to Visit 7
Measure: Mean (Standard Deviation); unit: seizures/month
Arm/Group | Placebo | Esl (BIA 2-093)
Number analyzed (Participants) | 129 | 134
seizures/month | 62.0 (186.19) | 36.6 (72.47)
Statistical Analysis 1: Comparison: Placebo vs Esl (BIA 2-093); Test type: Superiority or Other; p = 0.2490, ANCOVA

2. Primary Outcome: Responder Rate
Description: Responder rate defined as the number of patients with at least a 50% decrease in the standardised 4-week seizure frequency from the baseline period to the 12-week maintenance period.
Time Frame: baseline up to Visit 7
Measure: Number; unit: participants
Arm/Group | Placebo | Esl (BIA 2-093)
Number analyzed (Participants) | 129 | 134
participants | 40 | 41
Statistical Analysis 1: Comparison: Placebo vs Esl (BIA 2-093); Test type: Superiority or Other; p = 0.9017, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: from the time the patient gave informed consent until 14 days after the end of the follow-up period for Part I
Arm/Group | Placebo (Safety Set Part I) | Esl (Safety Set Part I)
Serious Adverse Events (participants affected / at risk) | 9/129 | 15/134
Other Adverse Events (participants affected / at risk) | 94/129 | 112/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Safety Set Part I) (N=129) | Esl (Safety Set Part I) (N=134)
VERTIGO (Ear and labyrinth disorders) | 0 | 1
COELIAC DISEASE (Gastrointestinal disorders) | 0 | 1
DEVICE MALFUNCTION (General disorders) | 0 | 2
DRUG WITHDRAWAL SYNDROME (General disorders) | 0 | 1
IRRITABILITY (General disorders) | 1 | 0
BRONCHOPNEUMONIA (Infections and infestations) | 0 | 2
INFECTIOUS MONONUCLEOSIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 3 | 1
VIRAL INFECTION (Infections and infestations) | 0 | 1
BRAIN HERNIATION (Injury, poisoning and procedural complications) | 0 | 1
BRAIN OEDEMA (Nervous system disorders) | 0 | 1
CONVULSION (Nervous system disorders) | 2 | 2
EPILEPSY (Nervous system disorders) | 0 | 1
GRAND MAL CONVULSION (Nervous system disorders) | 1 | 1
HYDROCEPHALUS (Nervous system disorders) | 1 | 0
HYPOTONIA (Nervous system disorders) | 1 | 0
PARTIAL SEIZURES WITH SECONDARY GENERALISATION (Nervous system disorders) | 0 | 1
STATUS EPILEPTICUS (Nervous system disorders) | 0 | 3
ASPHYXIA (Respiratory, thoracic and mediastinal disorders) | 1 | 0
VASCULAR PURPURA (Skin and subcutaneous tissue disorders) | 0 | 1
MEDICAL DEVICE CHANGE (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Safety Set Part I) (N=129) | Esl (Safety Set Part I) (N=134)
Headache (Nervous system disorders) | 8 | 18
Nasopharyngitis (Infections and infestations) | 45 | 15
Somnolence (Nervous system disorders) | 6 | 15
Convulsion (Nervous system disorders) | 14 | 13
Pyrexia (General disorders) | 7 | 10
Pharyngitis (Infections and infestations) | 9 | 9
Diplopia (Eye disorders) | 2 | 8
Vomiting (Gastrointestinal disorders) | 8 | 8
Nausea (Gastrointestinal disorders) | 1 | 7
Respiratory tract infection (Infections and infestations) | 7 | 7
Decreased appetite (Metabolism and nutrition disorders) | 1 | 6
Upper respiratory tract infection (Infections and infestations) | 5 | 6
Vertigo (Ear and labyrinth disorders) | 0 | 6
Viral infection (Infections and infestations) | 6 | 6
Agitation (Psychiatric disorders) | 1 | 5
Bronchitis (Infections and infestations) | 7 | 5
Dizziness (Nervous system disorders) | 2 | 5
Fatigue (General disorders) | 3 | 5
Viral upper respiratory tract infection (Infections and infestations) | 3 | 5
Weight increased (Investigations) | 2 | 5
Abdominal pain upper (Gastrointestinal disorders) | 0 | 4
Influenza (Infections and infestations) | 1 | 4
Rhinitis (Infections and infestations) | 7 | 4
Abdominal pain (Gastrointestinal disorders) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other